CLINICAL TRIAL: NCT03086096
Title: CIRSE Registry for LifePearl Microspheres
Acronym: CIREL
Status: Completed | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Responsible Party: Sponsor
Other Study IDs: 2
Record Dates: First submitted 2017-03-01; First posted 2017-03-22 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Carcinoma; Neoplasm Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LifePearl Microspheres loaded with Irinotecan — LifePearl Microspheres are embolisation microspheres for transcatheter chemoembolisation (TACE), that can be loaded with chemotherapeutic agents. In this registry, LifePearl Microspheres will be loaded with Irinotecan.

SUMMARY:
The application of transarterial chemoembolisation (TACE) using LifePearl Microspheres loaded with Irinotecan in liver-only or liver-dominant metastatic disease in patients with colorectal adenocarcinoma will be observed. The registry has the following objectives:

1. map the exact indications that the device is being used for and at which stage in treatment it is being applied
2. to assess observed treatment outcomes in terms of safety and effectiveness as well as trying to determine any predictive response factors

DETAILED DESCRIPTION:
CIREL will capture a broad spectrum of real clinical data on the delivery of transcatheter arterial chemoembolisation (TACE) using LifePearl Microspheres loaded with Irinotecan (LP-IRI) and the observed clinical outcomes. The aim of doing so is to improve our understanding of how LifePearl microspheres are administered as part of the standard treatment of colorectal adenocarcinoma with liver metastases in Europe. Ultimately, the collection of real-life data is intended to provide an evidence-base from which conclusions can be drawn on how to optimise treatment protocols and consequently the therapy outcome of TACE performed with LifePearl Microspheres.

The CIREL registry is a prospective multicentre observational (non-interventional) study. In order to meet the objective of collecting real-life data, all subjects receiving TACE with LifePearl Microspheres loaded with Irinotecan and fulfilling the inclusion criteria in all participating centres will be asked to participate. Patients are only asked to participate in the registry when they are treated with LifePearl Microspheres loaded with Irinotecan as part of the treatment determined by the treating clinician. In no way, will participation in the registry influence the way in which the patient is treated according to the treating clinician, or will it influence the quality of the treatment.

In order to measure changes in the quality of life of enrolled patients at different moments in time before and after treatment with LifePearl microspheres, CIREL will incorporate the EORTC QLQ-C30 questionnaire. The quality of life questionnaire is suggested to be offered to the patient at the following three points in time:

* Immediately (max. 1 week) before the treatment with LP-IRI
* 4-8 weeks after completion of the full treatment with LP-IRI
* 12-16 weeks after the completion of the full treatment with LP-IRI

Filling out the quality-of-life questionnaire is entirely voluntary for the patient. The patient will be offered to fill out the questionnaire in his/her mother tongue. The patient will have the choice to fill in the questionnaire either in hard copy or online via the electronic data capture system.

The CIREL registry will include central image analysis performed by the Fédération Francophone de Cancérologie Digestive (FFCD). The aim of the analyis is to detect possible associations between RECIST (v1.1) criteria and observed outcomes, reduce bias by providing a second reading and raise data quality.

The registry aims at enrolling up to 150 patients. The registry will stop enrolment two and a half years after the enrolment of the first patient, unless decided differently by the Steering Committee. Patients should be followed up until 65% of active patients are deceased and for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with liver-only or liver-dominant metastatic disease in patients with colorectal adenocarcinoma
* treatment with LifePearl Microspheres
* signed informed consent form
* 18 years or older

Exclusion Criteria:

* withdrawal of informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal adenocarcinoma and liver-only or liver-dominant metastatic disease
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Number of indications that the device is being used for, as assessed by stage and previous treatment(s) | 2.5 years
  The primary objective is to ultimately categorise observed usages as one of the following:
  * LifePearl as a first-line treatment
  * LifePearl as a consolidation or closing treatment with or without systemic therapy
  * Intensification of treatment with concomitant systemic therapy (objective: resectability and/or ablative therapy)
  * Salvage treatment in progressive patients pre-treated with systemic therapy, with or without concomitant systemic therapy
  * Combination treatment with ablation with a curative intent
  * Other

SECONDARY OUTCOMES:
Number of participants with acute and/or chronic adverse events according to CTCAE version 4.03. | 4 years
  Safety and Tolerability will be monitored during and after treatment with LP-IRI.
Time from observation until death due to any cause (or censoring) | 4 years
  Overall survival
Time from observation until disease progression or death | 4 years
  Progression-free survival (PFS) will be assessed by the investigator and central CT/MRI image analysis.
Time from observation until disease progression in the liver or death | 4 years
  Hepatic progression-free survival (liver-specific PFS) will be assessed by the investigator and central CT/MRI image analysis.
Proportion of patients with reduction in tumor burden, as assessed by RECIST (v.1.1) | 4 years
  Objective Tumour Response Rate will be assessed by the investigator and central CT/MRI image analysis.
Number of patients with tumour shrinkage at > 20% or >30% at first tumour assessment (4 - 8 wks) | 4 years
  Assessment of early tumour shrinkage serves as an early-on-treatment predictor of treatment efficacy.
Nadir of tumour response over the time of observation | 4 years
  Deepness of response (DpR) serves as a continuous measure, which defines the nadir of tumour response and serves as an early-on-treatment predictor of treatment efficacy.
Number of patients with secondary resections or ablative treatments following initial treatment with LP-IRI | 4 years
  Secondary resection/ablation
The quality of participants' lives, as assessed by the QLQ-C30 questionnaire (developed by EORTC) | 4 years
  Quality of Life questionnaires will be filled out:
  * Baseline: maximum 1 week before the first LP-IRI treatment
  * 2nd: 4-8 weeks after the whole LP-IRI treatment is completed
  * 3rd: 12-16 weeks after the whole LP-IRI treatment is completed

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Pereira, Prof., Study Chair — Interventional Radiologist at SLK Klinikum Heilbronn GmbH, Germany; Julien Taieb, Prof., Study Chair — Oncologist at Georges Pompidou European Hospital, Paris, France
Locations (1):
- CIRSE Cardiovascular and Interventional Radiological Society of Europe, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pereira PL, Iezzi R, Manfredi R, Carchesio F, Bansaghi Z, Brountzos E, Spiliopoulos S, Echevarria-Uraga JJ, Goncalves B, Inchingolo R, Nardella M, Pellerin O, Sousa M, Arnold D, de Baere T, Gomez F, Helmberger T, Maleux G, Prenen H, Sangro B, Zeka B, Kaufmann N, Taieb J. The CIREL Cohort: A Prospective Controlled Registry Studying the Real-Life Use of Irinotecan-Loaded Chemoembolisation in Colorectal Cancer Liver Metastases: Interim Analysis. Cardiovasc Intervent Radiol. 2021 Jan;44(1):50-62. doi: 10.1007/s00270-020-02646-8. Epub 2020 Sep 24. PMID 32974773
- [Derived] Pereira PL, Arnold D, de Baere T, Gomez F, Helmberger T, Iezzi R, Maleux G, Prenen H, Sangro B, Nordlund A, Zeka B, Bauer R, Kaufmann N, Pellerin O, Taieb J. A multicentre, international, observational study on transarterial chemoembolisation in colorectal cancer liver metastases: Design and rationale of CIREL. Dig Liver Dis. 2020 Aug;52(8):857-861. doi: 10.1016/j.dld.2020.05.051. Epub 2020 Jun 30. PMID 32620520